CLINICAL TRIAL: NCT06186830
Title: Validity, Reliability and Responsiveness of the Cognitive Exercise Therapy Approach Biopsychosocial Questionnaire in Individuals with Temporomandibular Disorder
Brief Title: Cognitive Exercise Therapy Approach Biopsychosocial Questionnaire (BETY-BQ) in Patient with Temporomandibular Disorders
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Collaborators: Karabuk University (Other)
Responsible Party: Principal Investigator, Harun Gençosmanoğlu, Principal Investigator, Karabuk University
Other Study IDs: 2023/1361
Record Dates: First submitted 2023-12-17; First posted 2024-01-02 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Temporomandibular Disorder; Temporomandibular Joint Disorders; Temporomandibular Joint Dysfunction Syndrome
Keywords: validity; reliability; responsiveness
MeSH Terms: conditions — Temporomandibular Joint Disorders; Temporomandibular Joint Dysfunction Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with temporomandibular disorder
  Interventions: Other: Validity and reliability analyses

INTERVENTIONS:
Other: Validity and reliability analyses — Validity and reliability analyses will be performed using Cognitive Exercise Therapy Approach Biopsychosocial Questionnaire, Patient Health Questionnaire-9, Patient Health Questionnaire-15, Generalized Anxiety Disorder-7, Short Form-36, Craniomandibular Pain and Disability Inventory, and Mandibular Function Impairment Questionnaire.

SUMMARY:
The aim of this study is to investigate the validity, reliability, and responsiveness of the Cognitive Exercise Therapy Approach-Biopsychosocial Questionnaire (BETY-BQ) in individuals with temporomandibular disorder. The following are alternative hypotheses of the study:

* BETY-BQ has significant convergence with the Patient Health Questionnaire-9 measuring depression.
* BETY-BQ has significant convergence with the Patient Health Questionnaire-15 measuring physical symptoms.
* BETY-BQ has significant convergence with the Generalized Anxiety Disorder-7 measuring anxiety.
* BETY-BQ has significant convergence with the Short Form-36 measuring quality of life.
* BETY-BQ has significant convergence with the Craniomandibular Pain and Disability Inventory measuring disability.
* BETY-BQ has significant convergence with the Mandibular Function Impairment Questionnaire measuring function.
* BETY-BQ has significant stability.
* BETY-BQ has significant internal consistency.

DETAILED DESCRIPTION:
Patient Health Questionnaire-9 (Depression), Patient Health Questionnaire-15 (Physical Symptoms), Generalized Anxiety Disorder-7 (Anxiety), Short Form-36 (Quality of Life), Craniomandibular Pain and Disability Inventory (Disability), and Mandibular Function Impairment Questionnaire (Function) will be administered to participants. For reliability analysis, test-retest stability evaluations will be repeated with the same questionnaire on 30 individuals with a 2-week interval. To determine responsiveness, the same questionnaire will be reapplied to the same 30 individuals at 3-month intervals.

ELIGIBILITY:
Inclusion Criteria:

* Having received a diagnosis of temporomandibular disorder

Exclusion Criteria:

* Experiencing difficulty in cooperating to fill out the questionnaires
* Being unwilling to participate in the study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with temporomandibular disorder
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-12-17 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Validity of BETY-BQ in measuring depression | Baseline
  Patient Health Questionnaire-9. Minimum and maximum values are 0 and 3 points, respectively. Higher scores mean a worse outcome.
Validity of BETY-BQ in measuring physical symptoms | Baseline
  Patient Health Questionnaire-15. Minimum and maximum values are 0 and 2 points, respectively. Higher scores mean a worse outcome.
Validity of BETY-BQ in measuring anxiety | Baseline
  Generalized Anxiety Disorder-7. Minimum and maximum values are 0 and 3 points, respectively. Higher scores mean a worse outcome.
Validity of BETY-BQ in measuring quality of life | Baseline
  Short Form-36. It is a 36-item valid and reliable evaluation with eight areas covering physical functioning, role limitations brought on by physical issues, bodily pain, general health perceptions, vitality, social functioning, role limitations brought on by emotional issues, and perceived mental health. The SF-36 also contains a single question called "health transition" that measures how respondents feel their over health status has changed over the course of a year.
Validity of BETY-BQ in measuring disability | Baseline
  Craniomandibular Pain and Disability Inventory. Minimum and maximum values are 0 and 3 points, respectively. Higher scores mean a worse outcome.
Validity of BETY-BQ in measuring function | Baseline
  Mandibular Function Impairment Questionnaire. Minimum and maximum values are 0 and 4 points, respectively. Higher scores mean a worse outcome.
Test-retest stability of BETY-BQ | From baseline to 2nd week
  The Cognitive Exercise Therapy Approach Biopsychosocial Questionnaire will be repeated on 30 individuals with a 2-week interval.
Internal consistency of BETY-BQ | Baseline
  Cognitive Exercise Therapy Approach Biopsychosocial Questionnaire. Minimum and maximum values are 0 and 4 points, respectively. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Harun Gençosmanoğlu, PT, MSc, Principal Investigator — Karabük University
Locations (2):
- Turkey (Türkiye) (2):
  - Karabük University, Karabük, Karabük Province
  - Hacettepe University, Ankara

IPD SHARING:
Plan to Share IPD: No